CLINICAL TRIAL: NCT00150527
Title: Specific Effects of Escitalopram on Neuroendocrine Response
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Dr. Nicholas Delva, Dalhousie University
Other Study IDs: ESCIT001
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: antidepressive agents
MeSH Terms: interventions — Citalopram; Escitalopram; Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Citalopram — 40 mg, pill, single dose
  Other Names: Celexa
Drug: Escitalopram — 20 mg, pill, single dose
Drug: Dexamethasone — 1 mg, pill, single dose
Behavioral: Cold Pressor Test — single test

SUMMARY:
Citalopram, a selective serotonin reuptake inhibitor (SSRI), is used as a neuroendocrine probe in human subjects to assess serotonin (5-hydroxytryptamine; 5-HT) function as reflected in prolactin and plasma cortisol release. Citalopram is a racemic mixture of equal parts of the S(+) and R(-) enantiomers. The S(+) form ("escitalopram") has been identified as being the active isomer and inhibitor of serotonin reuptake and consequently antidepressant activity is associated almost exclusively with the S-enantiomer. Escitalopram has been shown to be approximately twice as potent as citalopram at the primary, high-affinity binding site on the human serotonin transporter. Interestingly, investigations have suggested an antagonistic interaction of the R- and S-enantiomer at an allosteric binding site on the serotonin transporter. This antagonism has been shown in animal studies where the addition of R-citalopram to escitalopram treatments significantly counteracts the antidepressant and anti-anxiolytic effects of escitalopram. From these clinical and experimental data, the researchers can anticipate that escitalopram would increase cortisol and prolactin in the neuroendocrine challenge paradigm more effectively than citalopram.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* The age range will be restricted to between 18 and 59 years of age.
* Subjects must be fit and have no history of significant illness.
* Subjects must have no risk factors for HIV or viral hepatitis.
* Subjects must be non-smokers, free of medication, and consume alcoholic and caffeinated beverages in moderation.
* Subjects must also be in good psychological health with no history of psychiatric illness.

Exclusion Criteria:

* Personal history of psychiatric illness, habitual smoking, illicit or prescription drug use, high intake of alcohol (>10 drinks/week) or caffeine (>500 mg caffeine/day), shift work, pregnancy, personal or familial history of seizures, significant medical illness or treatment in the last six months, significant physical or laboratory abnormalities, or current use of a weight loss diet.
* Women entering the study must be on a reliable form of birth control, i.e., tubal ligation, hysterectomy, oral contraceptives, abstinence, or vasectomy in partner.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal healthy people
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2005-09; Primary Completion 2006-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The effect of the drugs on serum cortisol and ACTH following a single dose of each drug. | 4hrs

SECONDARY OUTCOMES:
Side effects following a single dose of the drug | 4hrs

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Delva, MD, Principal Investigator — Queen's University
Locations (1):
- Providence Centre, Mental Health Services, Kingston, Ontario, Canada